CLINICAL TRIAL: NCT06231394
Title: Effectiveness of Multimodal Pelvic Floor Rehabilitation Program in Children With Different Types of Urinary Incontinence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Damla Korkmaz Dayican (Other)
Collaborators: Biruni University (Other); Dokuz Eylul University (Other)
Responsible Party: Sponsor-Investigator, Damla Korkmaz Dayican, Lecturer, Izmir Tinaztepe University
Organization: Izmir Tinaztepe University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: T-DAYICAN-001
Record Dates: First submitted 2024-01-18; First posted 2024-01-30 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Urinary Incontinence; Nocturnal Enuresis; Daytime Wetting; Pelvic Floor Disorders; Children, Only; Pediatric Disorder
Keywords: urinary incontinence; nocturnal enuresis; daytime incontinence; pediatric; pelvic floor rehabilitation
MeSH Terms: conditions — Urinary Incontinence; Nocturnal Enuresis; Diurnal Enuresis; Pelvic Floor Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- daytime incontinence (Active Comparator): This group will consist of participants who will be diagnosed with daytime incontinence by a pediatric urologist according to the International Children's Continence Society criteria.
  Interventions: Other: multimodal pelvic floor rehabilitation
- nocturnal enuresis (Active Comparator): This group will consist of participants who will be diagnosed with nocturnal enuresis by a pediatric urologist according to the International Children's Continence Society criteria.
  Interventions: Other: multimodal pelvic floor rehabilitation
- combined daytime incontinence and nocturnal enuresis (Active Comparator): This group will consist of participants who will be diagnosed with combined daytime incontinence and nocturnal enuresis by a pediatric urologist according to the International Children's Continence Society criteria.
  Interventions: Other: multimodal pelvic floor rehabilitation

INTERVENTIONS:
Other: multimodal pelvic floor rehabilitation — A multimodal pelvic floor rehabilitation program will be performed on all children for 10 weeks, two days a week and approximately 45 minutes. A multimodal pelvic floor rehabilitation will include education, bladder and bowel training, manual techniques, exercise training (diaphragmatic breathing exercise, pelvic floor muscle training, trunk stabilization exercises based on developmental kinesiology) and a home program. The home program will be given on other days of the week.

SUMMARY:
Urinary incontinence is defined by the International Children's Continence Society as involuntary urinary leakage that can be continuous or intermittent in children aged five and over. Urinary incontinence is divided into subgroups of daytime incontinence, nocturnal enuresis and combined daytime incontinence and nocturnal enuresis. Different pelvic floor rehabilitation programs appear to be effective in children with daytime incontinence and nocturnal enuresis but mostly focus on the pelvic floor muscle training component. However, pelvic floor rehabilitation includes many components such as education, lifestyle changes, manual techniques, pelvic floor muscle training, functional exercises, biofeedback therapy, electrical stimulation and home program. However, there is no study examining the effectiveness of a multimodal pelvic floor rehabilitation program in the treatment of children with urinary incontinence. It is also unclear for which urinary incontinence type the multimodal pelvic floor rehabilitation program will be more effective. Therefore, investigators aim to compare the effects of a multimodal pelvic floor rehabilitation program on lower urinary tract symptoms, pelvic floor muscles and other related muscle functions in children with different urinary incontinence types. Children between the ages of 5 and 18 who were diagnosed with urinary incontinence by applying to Ege University Faculty of Medicine, Department of Pediatric Urology will be included in the study. Participants will be divided into three groups: daytime incontinence, nocturnal enuresis, and combined daytime incontinence and nocturnal enuresis. A multimodal pelvic floor rehabilitation program will be performed on all children for 10 weeks, two days a week and approximately 45 minutes. A multimodal pelvic floor rehabilitation program will include education, bladder and bowel training, manual techniques, exercise training (diaphragmatic breathing exercise, pelvic floor muscle training, trunk stabilization exercises based on developmental kinesiology) and a home program. Children's lower urinary symptoms will be assessed with the Dysfunctional Voiding and Incontinence Scoring System, Bladder and Bowel Dysfunction Questionnaire, Childhood Bladder and Bowel Dysfunction Questionnaire, bladder and bowel diary, and the functions of the pelvic floor muscles and other related muscles will be assessed with superficial electromyography and ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 5-18
* Having been diagnosed with urinary incontinence according to the International Children's Continence Society criteria by a pediatric urologist (daytime incontinence, nocturnal enuresis, combined daytime incontinence and nocturnal enuresis)
* Signed the informed consent form
* Parent or child's ability to read and write Turkish

Exclusion Criteria:

* Presence of neurogenic lower urinary tract dysfunction
* Presence of anatomical changes and malformations in the urinary system
* Presence of active urinary system infection
* Having previously undergone surgery to treat urinary incontinence
* The child has any condition that would prevent participation in assessment or treatment (cognitive impairment, mental retardation, orthopedic disease or surgery, etc.)
* Presence of congenital thorax deformity
* The child has received pelvic floor rehabilitation within the last six months

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Dysfunctional Voiding and Incontinence Scoring System (DVAISS) | pre-intervention; immediately after the intervention
  DVAISS was developed to evaluate the severity of dysfunctional voiding and incontinence symptoms by Akbal et al. DVAISS consists of 14 questions examining daytime and nighttime symptoms, bladder and bowel habits, and quality of life. DVAISS score is based on the estimated odds ratio for each question between participants and controls. If the estimated odds ratio of the question is between 2 and 10, one point is given and if the estimated odds ratio is greater than 50, five points are given. The total score varies between 0 and 35. The increase in the total score indicates that the severity of the symptoms increases. A score of 8.5 or higher on the scale indicates the presence of bladder and bowel dysfunction. The Cronbach Alpha value of the scale was determined as 0.50.
Bladder and Bowel Dysfunction Questionnaire (BBDQ) | pre-intervention; immediately after the intervention
  BBDQ was developed to evaluate symptoms of bladder and bowel dysfunction by Afshar et al. The Turkish validity and reliability was conducted by Kaya Narter et al. BBDQ includes 13 questions about bladder and bowel symptoms such as incontinence, voiding, enuresis, dysuria, and constipation. Each question is scored on a 5-point Likert scale ranging from zero to four points. The total score varies between 0 and 52. As the total score increases, symptom severity worsens. A score of 11 points or above is considered bladder and bowel dysfunction. Cronbach Alpha value of the scale was found to be 0.727.
Childhood Bladder and Bowel Dysfunction Questionnaire (CBBDQ) | pre-intervention; immediately after the intervention
  CBBDQ consists of a total of 18 questions that assess bladder and bowel symptoms in children. CBBDQ has two subdimensions: Bladder Symptoms Scale (10 questions) and Bowel Symptoms Scale (8 questions). Considering the presence of children's symptoms in the last month, CBBDQ is filled out by parents on a 5-point Likert scale ranging from zero (no symptoms) to four points (symptoms occur almost every day). The total score from the scale varies between 0 and 72. As the total score increases, symptoms worsen. The Turkish validity and reliability of the scale was conducted by Aydin et al. Cronbach Alpha values were determined as 0.74 and 0.71 for bladder and bowel subdimensions, respectively.
Bladder Diary | pre-intervention; immediately after the intervention
  The bladder diary is a simple and non-invasive method that objectively assesses bladder habits. The bladder diary is used to record the type and amount of consumed fluid over 48 hours, the amount and duration of urination, urgency, urinary frequency, and the amount and time of urinary incontinence. The bladder diary is desirable to record for two consecutive days. The amount of consumed fluid and the urination is expressed in milliliters (ml), and the duration of urination is expressed in seconds (sec).
Bowel Diary | pre-intervention; immediately after the intervention
  The ICCS recommends the use of a seven-day bowel diary in children with lower urinary tract symptoms due to the close relationship between bladder and bowel function. The bowel diary questions the defecation frequency, pain during defecation, urgency, stool type, and the presence of fecal incontinence. The Bristol Stool Scale is used for stool type. The bowel diary consists of seven pictures and stool form descriptors and allows children to express participants' bowel movement intensity.

SECONDARY OUTCOMES:
Superficial Electromyography (EMG) | pre-intervention; immediately after the intervention
  A NeuroTrac MyoPlus 4 PRO (Verity Medical LTD., UK) type EMG device will be used in the study. Bioelectrical activities of the muscles (pelvic floor muscles, abdominal muscles, diaphragm, multifidus) will be recorded with disposable 3.2 x 3.2 cm superficial electrodes. To reduce skin impedance, the skin area will be cleaned with an alcohol swab. Active electrodes will be placed on the right side of the body, parallel to the muscle fibers, according to the reference points. The reference electrode will be placed on the anterior superior iliac spine. Measurements will be performed during five seconds of maximal voluntary contraction ('work' phase EMG activity) and five seconds of relaxation ('rest' phase EMG activity) of the pelvic floor muscles. Measurements will be repeated for three times. The graphic and numerical data provided by the device will be recorded in the evaluation form.
Ultrasonography (USG) | pre-intervention; immediately after the intervention
  Pelvic floor displacement, endurance, phasic contraction and coordination, bladder volume, bladder wall thickness and post voiding residue, abdominal muscles and multifidus thicknesses, diaphragmatic displacement and thickness will be measured. A transabdominal diagnostic USG device (Sonospace SSI-600) with a low frequency (2-5 MHz) curvilinear transducer will be used. Muscle thickness and distance measurements will be made during frozen imaging. Muscle thickness will be measured between the upper border of the muscle fascia, which appears as a white line, and the end point of the lower border. Measurements will be taken at the expiration and during a five-second pelvic floor muscle contraction. Both measurement results will be recorded in millimeters. All measurements will be repeated three times and the average values will be noted on the evaluation form.

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Razak Özdinçler, Study Director — Fenerbahçe University; Damla Korkmaz Dayıcan, Principal Investigator — İzmir Tınaztepe University; Özge Çeliker Tosun, Principal Investigator — Dokuz Eylul University; Büşra Palaz, Principal Investigator — Dokuz Eylul University; İbrahim Ulman, Principal Investigator — Ege University; Ali Tekin, Principal Investigator — Ege University; Sibel Tiryaki, Principal Investigator — Ege University
Locations (1):
- Ege University Faculty of Medicine, Department of Pediatric Urology, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No